CLINICAL TRIAL: NCT03180164
Title: Anxiety and Depression in Chronic Airways Diseases
Brief Title: Depression in Chronic Airways Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, fareda ahmed mohamed, principle investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CLD
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Chronic Lung Disease
MeSH Terms: interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chronic lung diseases (Other): bronchiectasis , bronchial asthma and chronic obstructive pulmonary disease assess anxiety and depression by hospital anxiety and depression scale
  Interventions: Other: hospital anxiety and depression scale

INTERVENTIONS:
Other: hospital anxiety and depression scale — self-assessment scale has been developed and found to be a reliable instrument for detecting states of depression and anxiety in the setting of an hospital medical outpatient clinic

SUMMARY:
Chronic airways diseases involve alterations in the person's social roles, relationships and self-perception so demands continual psychological adjustment .

Also Kunik studied patients with chronic breathing disorders for depression and anxiety and found that 65% of patients were positive for depression and anxiety.

Shackell found that patients' anxiety and fears of breathlessness and dying extended into the night and were aggravated by feelings of isolation and frustration. One patient reported that they often thought 'am I going to see the next morning?'

DETAILED DESCRIPTION:
This fear and sense of helplessness can lead to panic and evidence suggests that patients with chronic breathlessness often call for emergency assistance during the night According to GOLD report 2017, anxiety and depression in chronic obstructive pulmonary disease patients are both associated with poor prognosis.

Much of the evidence explored so far relates to chronic obstructive pulmonary disease. While other chronic lung diseases have received less attention In addition to, several studies have been found relationship between asthma and psychological disturbance .One review of literature describes an increased prevalence of psychological co-morbidity in asthmatic adults and another research suggests that anxiety and depression are more common in patients with moderate to severe asthma than in the general population Gift. found significantly greater self-reported depression scores among patients with chronic obstructive pulmonary disease receiving prednisone compared to patients not receiving any steroids.

Interestingly, the psychiatric sequel of steroid treatment are often sudden in onset and appear to generally occur within 2 weeks after steroid introduction

ELIGIBILITY:
Inclusion Criteria:

* Chronic airways diseases as chronic obstructive pulmonary disease, bronchial asthma, bronchiectasis

Exclusion Criteria:

* Diabetes Mellitus and Hypertension.
* Cardiac diseases.
* Chronic renal and liver diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
compare anxiety and depression in different forms of chronic lung diseases | 10 minutes
  by hospital anxiety and depression scale

CONTACTS AND LOCATIONS:
Overall Officials: Reham Mohamed El-Morshedy, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: No